CLINICAL TRIAL: NCT00484497
Title: A Randomized, Double-Blind, Placebo-Controlled Trial for the Evaluation of a Food Supplement on Sleep Quality in Primary Insomnia Patient
Brief Title: Evaluation of a Food Supplement on Sleep Quality
Acronym: Cyclamax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Persee Medica (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGS2006/0492
Record Dates: First submitted 2007-06-01; First posted 2007-06-11 (Estimated); Last update posted 2007-06-11 (Estimated); Status verified 2007-06

CONDITIONS: Insomnia
Keywords: Sleep quality; food supplement; randomized controlled trial; actigraphy; Leeds; Volunteers presenting moderate primary insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cyclamax

SUMMARY:
The purpose of this study is to evaluate the efficacy on sleep quality of a food supplement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged between 25 to 65 years
* Patient diagnosed for primary Insomnia (threshold for inclusion: 10 on the ISI scale)
* Healthy volunteer without diurnal sleep (total score for inclusion must be less than 10 on the Epworth scale)
* Patient affiliated to the French Social Security
* Patient who gave written informed consent

Exclusion Criteria:

* Secondary insomnia
* History of severe psychiatric disorder, assessed by the MINI test
* Resistance to Hypnotic drugs
* Anxiety, depression, suicide, detected by the Beck Depression Inventory
* Acute Pathology during the precedent three years
* Breast feeding and pregnancy women
* Non compliant volunteer
* Hypersensibility to treatment composant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Sleep quality assessed by the Leed Sleep Evaluation Questionnaire, measured after one month of treatment

SECONDARY OUTCOMES:
Sleep quality assessed by the Leed Sleep Evaluation - Questionnaire, measured 15 days after treatment withdrawal
Sleep quality assessed by a Sleep diary completed each day during all the study period by the participants
Sleep efficiency measured by ambulatory actigraphy (2 period)
Evolution of melatonin/6sulfatoxymelatonin ratio (before and after treatment)
Clinical General Impression of the clinician, before and after treatment.
Safety of the treatment (adverse event reporting)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cornu, MD, Principal Investigator — Clinical Research Center
Locations (1):
- Clinical Research Center- Hopital Cardiologique, Lyon, France

REFERENCES:
- [Derived] Cornu C, Remontet L, Noel-Baron F, Nicolas A, Feugier-Favier N, Roy P, Claustrat B, Saadatian-Elahi M, Kassai B. A dietary supplement to improve the quality of sleep: a randomized placebo controlled trial. BMC Complement Altern Med. 2010 Jun 22;10:29. doi: 10.1186/1472-6882-10-29. PMID 20569455